CLINICAL TRIAL: NCT07045285
Title: Prospective Randomized Trial Comparing Outcomes Of Episiorrhaphy Using Vicryl Rapid Coated 2/0 Versus Vicryl 2/0 Plus Triclosan
Brief Title: Prospective Randomized Trial On Episiorrhaphy
Acronym: VICRYL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Valeria Maria Savasi, Professor, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: VICRYL
Record Dates: First submitted 2025-05-02; First posted 2025-07-01 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Suture Materials
Keywords: Episiotomy; pregnancy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- antibacterial sutures (Experimental): antibacterial Vicryl Plus 2/0 sutures.
  Interventions: Device: Antibacterial Vicryl Plus 2/0
- non-antibacterial sutures (Active Comparator): standard (non-antibacterial) Vicryl 2/0 sutures.
  Interventions: Device: Standard Vicryl 2/0

INTERVENTIONS:
Device: Antibacterial Vicryl Plus 2/0 — antibacterial Vicryl Plus 2/0 sutures are multifilament absorbable synthetic sutures that are coated with triclosan, a purified antimicrobial.
  Arms: antibacterial sutures
Device: Standard Vicryl 2/0 — Vicryl rapid coated 2/0 sutures are multifilament absorbable synthetic sutures not treated with any antimicrobial.
  Arms: non-antibacterial sutures

SUMMARY:
An episiotomy refers to the incision of the perineum performed to increase the space of the vaginal opening to facilitate the birth of the newborn. Subsequently, the incision is closed by aligning the tissues without cutaneous and vascular alterations. Although a systematic review and metanalysis demonstrated that sutures coated with triclosan, a purified antimicrobial, prevent surgical site infections, there is no evidence in the literature regarding the use of antibacterial sutures for perineal plane compared to standard ones.

Therefore, the goal of this clinical trial is to compare the outcomes of incisions performed with standard Vicryl 2/0 sutures and antibacterial Vicryl Plus 2/0 sutures.

The study involves women giving birth at the Vittore Buzzi Children's Hospital, for whom an incision is necessary at the time of delivery. Participants will be evaluated at 48 hours (at the time of the hospital discharge visit), 40 days (at the postpartum visit), and 6 months (by phone interview) after delivery.

In particular, the aim of this study is to assess whether:

* antibacterial Vicryl Plus 2/0 sutures reduce pain after delivery;
* antibacterial Vicryl Plus 2/0 sutures improve the overall wound healing rate, avoid sexual, urinary or bowel disorders and the need for additional pharmacological, surgical, or physiotherapeutic interventions (in case of suboptimal wound healing).

This study also aims to validate a new ASEPSIS ( Additional Treatment, Serous exudate, Erythema, Purulent exudate, Separation of deep tissues, Isolation of bacteria and Stay) score for the evaluation of healing outcomes of episiotomies.

This is a double-blind, parallel-group randomized controlled trial. After obtaining informed consent, participants are randomly assigned either to the experimental group or the control group. Participants do not know the group they belong to, as the researchers; only the healthcare professional performing the suture knows it.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at term (more than 37 weeks);
* age between 18 and 40 years;
* women who give consent to participate in the study;
* women who give birth during the recruitment period;
* women for whom an episiotomy is necessary at the time of delivery.

Exclusion Criteria:

* age lower than 18 years and more than 40 years;
* gestational age lower than 37 weeks;
* diabetes mellitus or gestational diabetes;
* African and South-East Asian ethnicities;
* cigarette smoking;
* BMI higher than 30;
* anemia;
* lack of consent to participate;
* complicated episiotomy and/or presence of other spontaneous perineal lacerations;
* women lost to follow-up or who have undergone non-gynecological perineal interventions during the follow-up period.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Pain evaluation | 48 hours, 40 days and six months postpartum.
  Pain is defined through a Swab test (based on a pain scale known as the Visual Analogue scale (VAS) with a score from 0 to 10 (0= no pain, 10=worst imaginable pain)

SECONDARY OUTCOMES:
Re-suturing | at 48 hours and 40 days after delivery
  Re-suturing (performed or not performed)
Wound Healing Status Assessed by ASEPSIS Score | 48 hours, 40 days and six months postpartum.
  The ASEPSIS (Additional treatment, Serous exudate, Erythema, Purulent exudate, Separation of deep tissues, Isolation of bacteria, and Stay) score evaluates the extent of wound healing complications after delivery. It quantifies serous exudate, erythema, purulent exudate, and wound dehiscence on the suture line. Additional points are assigned for antibiotic use, drainage of purulent material, bacterial isolation from cultures, and hospitalization exceeding 14 days. Scores range from 0 to over 40, with higher scores indicating more severe wound infection or healing disturbance.
Functional disorders secondary to episiotomy repair | Assessed at 6 months postpartum
  Assessment of dyspareunia (present or absent), urinary disorders (present or absent) ,and bowel disorders (present or absent)

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Savasi, MD, PhD, Principal Investigator — ASST Fatebenefratelli Sacco
Locations (1):
- Ospedale dei Bambini "Vittore Buzzi", Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No